CLINICAL TRIAL: NCT01830569
Title: Feasibility and Impact of an Evidence-based Electronic Decision Support System on Diabetes Care in Family Medicine: a Cluster Randomized Controlled Trial
Brief Title: Impact of an Evidence-based Electronic Decision Support System on Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Bert Aertgeerts, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S55183
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Decision Support Systems, Clinical; Evidence-Based practice; Family Practice
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBMeDS group (Experimental): The regular Evidence Linker and the EBMeDS system will be available in this group.
  Interventions: Behavioral: The EBMeDS system; Other: Evidence Linker
- Control group (Other): The regular Evidence Linker will be available in this group.
  Interventions: Other: Evidence Linker

INTERVENTIONS:
Behavioral: The EBMeDS system — The EBMeDS system receives structured patient data from the electronic medical records in HealthOne and returns reminders, therapeutic suggestions and diagnosis-specific links to guidelines. Electronic forms and calculators (e.g. a calculator for glomerular filtration) are integrated in the system.
  The original EBMeDS system was developed by Duodecim in Finland and covers a full spectrum of all clinical areas. Relevant reminders in all clinical areas are shown to the physicians in the intervention group.
  Arms: EBMeDS group
Other: Evidence Linker — The Evidence Linker is already integrated in Belgian routine practice since 2012 and could be considered as part of the usual care process. When entering a diagnosis coded in ICPC, relevant clinical practice guidelines are retrieved by the Evidence Linker and could by consulted on the initiative of the family physician.

SUMMARY:
The purpose of this study is to assess the feasibility of the use of an evidence-based decision support system (EBMeDS) in daily Belgian family medicine and to study the effectiveness of EBMeDS use on improving diabetes care.

DETAILED DESCRIPTION:
The purpose of this study is to assess the feasibility of the use of an evidence-based decision support system (EBMeDS) in daily Belgian family medicine and to study the effectiveness of EBMeDS use on improving diabetes care.

Specific research questions are:

* Does family physicians use the EBMeDS system in daily practice?
* Does the use of the EBMeDS system by family physicians leads to an improvement in diabetes control compared to the control group?

ELIGIBILITY:
Inclusion Criteria:

* Patients are 18 years or older.
* Patients have their electronic medical records registered by one of the included family physicians. Medical records are not centralized in Belgium. Patients are free to choose any physician, and can even see several physicians at the same time. To encourage a patient to have their medical records held by a single physician, 'Global Medical Records' werr introduced a decade ago. In return for a registration fee, patients can choose a main general practitioner who keeps their central medical records. This registration is a requirement for patient inclusion in the trial. Patients with 'Global Medical Records' are reimbursed a larger proportion of the consultation fees by the health insurance fund.
* Patients have an established diagnosis of diabetes at the baseline time point of the study (identified as having (1) an ICPC (International Classification of Primary Care) code of diabetes or (2) a prescription for a diabetes-specific or (3) the necessary labo results to confirm diabetes)

Exclusion Criteria:

* Pregnancy
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Pre- to post-implementation change in HbA1c. | Outcome will be collected at five points in time: before the start of the study, at 3 months, at 6 months, at 9 months and at 12 months

SECONDARY OUTCOMES:
Pre- to post-implementation change in cholesterol levels. | Outcome will be collected at five points in time: before the start of the study, at 3 months, at 6 months, at 9 months and at 12 months
Pre- to post-implementation change in blood pressure measurements. | Outcome will be collected at five points in time: before the start of the study, at 3 months, at 6 months, at 9 months and at 12 months
Pre- to post-implementation change in a composite patient score. | Outcome will be collected at five points in time: before the start of the study, at 3 months, at 6 months, at 9 months and at 12 months
  The composite patient score consists of reaching the evidence-based targets for glycated hemoglobin, blood pressure (systolic and diastolic) and cholesterol. Differences between pre- and post-implementation will be forming the outcomes scores.
Pre- to post-implementation change in a composite process score. | Outcome will be collected at five points in time: before the start of the study, at 3 months, at 6 months, at 9 months and at 12 months
  The process composite score consists of meeting the evidence-based targets of the number of blood pressure measurements, the number of laboratory results of HbA1c, cholesterol and micro-albuminuria, a prescription of statin (yes/no), if high cardiovascular risk a prescription of aspirin/clopidogrel (yes/no), if hypertension or nephropathy ACE inhibition/sartan (yes/no). Differences between pre- and post-implementation will be forming the outcomes scores.

OTHER OUTCOMES:
Actual use of the EBMeDS system | Outcomes will be collected at five points in time: before the start of the study, at 3 months, at 6 months, at 9 months and at 12 months
  Scripts are automatically triggered, users can see that a script is available from their main screen but have to click before seeing the script content. As such, click events can give an indication of physicians' interest to use the system. Following data of actual use are collected in the log file: the percentage of triggered scripts that are opened, the type of scripts that are opened (reminder, interaction, contraindication, drugs to avoid, indication or GuidelineLink), the number of requests to open the details of the script or the script information.

CONTACTS AND LOCATIONS:
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Heselmans A, Delvaux N, Laenen A, Van de Velde S, Ramaekers D, Kunnamo I, Aertgeerts B. Computerized clinical decision support system for diabetes in primary care does not improve quality of care: a cluster-randomized controlled trial. Implement Sci. 2020 Jan 7;15(1):5. doi: 10.1186/s13012-019-0955-6. PMID 31910877
- [Derived] Heselmans A, Van de Velde S, Ramaekers D, Vander Stichele R, Aertgeerts B. Feasibility and impact of an evidence-based electronic decision support system for diabetes care in family medicine: protocol for a cluster randomized controlled trial. Implement Sci. 2013 Aug 5;8:83. doi: 10.1186/1748-5908-8-83. PMID 23915250